CLINICAL TRIAL: NCT07065331
Title: A Phase I, Open-label, Single-dose Study to Evaluate the Pharmacokinetics of Inhaled AZD8630 in Adolescents With Asthma
Brief Title: A Study of Inhaled AZD8630 in Adolescents With Asthma
Acronym: APkITA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D6830C00005
Record Dates: First submitted 2025-06-11; First posted 2025-07-15 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Asthma
Keywords: Dry powder inhaler; Anti-Thymic stromal lymphopoietin
MeSH Terms: conditions — Asthma | interventions — Dry Powder Inhalers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- AZD8630 (Experimental): Participants will receive single inhaled dose of AZD8630 on Day 1 via dry powder inhaler.
  Interventions: Drug: AZD8630; Device: Dry powder inhaler

INTERVENTIONS:
Drug: AZD8630 — Single inhaled dose of AZD8630 via dry powder inhaler.
Device: Dry powder inhaler — Single inhaled dose of AZD8630 via dry powder inhaler.

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic (PK) profile, safety, tolerability, and immunogenicity of single inhaled dose of AZD8630 administered in adolescent participants with asthma as well as the safety and performance of the dry powder inhaler.

DETAILED DESCRIPTION:
This is a Phase 1, open label, single dose study that will be conducted in adolescent participants with asthma where the participants will receive AZD8630 administered via dry powder inhaler.

The study will be comprised of:

* A screening period.
* A treatment period.
* A post treatment period.
* A final Follow-up visit.

ELIGIBILITY:
Key Inclusion Criteria:

* Physician prescribed daily use of asthma medication.
* Pre-bronchodilator Forced expiratory volume in one second (FEV1) ≥ 50% of the predicted normal value.
* Asthma control questionnaire-5 (ACQ-5) < 1.5 at Screening and Study Day 1.

Key Exclusion Criteria:

* History of any clinically important disease or disorder.
* History of any chronic respiratory disorders (except asthma).
* Acute exacerbation of asthma within 4 weeks of Screening.
* Life -threatening asthma.
* Completed treatment for respiratory infection with antibiotics within 4 weeks of Screening.
* History of acquired or inherited immunodeficiency disorders.
* Oral immunotherapy, including stable maintenance dose allergen-specific oral immunotherapy.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2025-06-11 (Actual); Primary Completion 2025-09-19 (Actual); Study Completion 2025-09-19 (Actual)

PRIMARY OUTCOMES:
Area under the serum concentration-time curve from time zero to 24 hours (AUC0-24) | Up to Day 9
  The AUC0-24 of AZD8630 after administered as single inhaled dose in adolescent participants with asthma will be evaluated.
Maximum observed drug concentration (Cmax) | Up to Day 9
  The Cmax of AZD8630 after administered as single inhaled dose in adolescent participants with asthma will be evaluated.
Time to reach peak or maximum observed concentration (Tmax) | Up to Day 9
  The Tmax of AZD8630 after administered as single inhaled dose in adolescent participants with asthma will be evaluated.

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | From screening until Follow-up (Day 9)
  The safety and the tolerability of AZD8630 in adolescent participants with asthma will be evaluated.
Incidences of anti-drug antibodies (ADA) of AZD8630 | Day 1 and Day 9
  The immunogenicity of AZD8630 in adolescent participants with asthma will be evaluated.
Number of participants with AEs associated with dry powder inhaler | Day 1
  The safety and the performance of the dry powder inhaler device in adolescent participants with asthma will be evaluated.
Number of participants with dry powder inhaler deficiencies | Day 1
  The safety and the performance of the dry powder inhaler in adolescent participants with asthma will be evaluated.
Number of participants with dose administration confirmation | Day 1
  The safety and the performance of the dry powder inhaler in adolescent participants with asthma will be evaluated.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Research Site, Bakersfield, California
  - Research Site, Miami Lakes, Florida
  - Research Site, Lafayette, Louisiana
  - Research Site, Raleigh, North Carolina
  - Research Site, Toledo, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Spartanburg, South Carolina
  - Research Site, Boerne, Texas
  - Research Site, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secureresearchenvironmentVivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/